CLINICAL TRIAL: NCT04622852
Title: Are Pegs Better Than Screw for Osteofixation of Proximal Humeral Fractures?
Brief Title: Pegs for Osteofixation of Proximal Humeral Fractures
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tore Fjalestad, MD. PhD. Senior Consultant Ortophaedic Surgeon, Oslo University Hospital
Other Study IDs: 2017/681
Record Dates: First submitted 2020-11-03; First posted 2020-11-10 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Implant Complication; Proximal Humeral Fracture; Avascular Necrosis of Humerus
Keywords: Humeral head; Screw penetration; Peg penetration; Avascular necrosis
MeSH Terms: conditions — Shoulder Fractures; Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: ALPS-PHP device: Patients operated with angular stable plate for displaced PHF with an ALPS plate
  Interventions: Device: Open reduction internal fixation (ORIF) with an angular stable plate
- Group B: Philos device: Patients operated with angular stable plate for displaced PHF with a Philos plate
  Interventions: Device: Open reduction internal fixation (ORIF) with an angular stable plate

INTERVENTIONS:
Device: Open reduction internal fixation (ORIF) with an angular stable plate — Operative treatment of proximal humeral fracture

SUMMARY:
Patients treated operative for Proximal humeral fractures with angular stable device (Philos plate or ALPS-PHP)

DETAILED DESCRIPTION:
From a cohort of patients treated for displaced Proximal humeral fractures (PHF) in the period July 2017 - August 2019 patients with the 11-B2 and 11-C2 PHF according to AO/OTA 2007 fracture classification were selected according to age and gender to be compared with patients operated with a Philos plate within the same fracture group, age and gender to be matched for adverse events:

1. Radiographic evidence of penetration of pegs (ALPS-PHP) or screws (Philos) into the glenohumeral joint (primary outcome) and
2. Avascular head necrosis / sinking / need of re-surgery
3. Clinical PROMS

ELIGIBILITY:
Inclusion Criterion:

* Acute proximal humeral fracture
* AO/OTA type 11-B2 or 11C2

Exclusion Criteria:

* Not eligible to surgical treatment
* Non-compliant
* Former shoulder fracture or symptomatic shoulder illness
* Drug abuser

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with an acute PHF for surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Peg penetration into glenohumeral joint | 12 months
  Radiographic or CT verified peg penetration
Screw penetration into glenohumeral joint | 12 months
  Radiographic or CT verified screw penetration

SECONDARY OUTCOMES:
Humeral head deformation | 12 months
  Avascular head necrosis or Sinking
Shoulder function | 12 months
  Constant-Murley score
Self reported shoulder function | 12 months
  Oxford scoulder score
Quality of life | 12 months
  Generic 15D score

CONTACTS AND LOCATIONS:
Overall Officials: Tore Fjalestad, MD, PhD., Principal Investigator — Oslo University Hospital, Ortophaedic Dept.
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
No plan has been decided

REFERENCES:
- [Derived] Bones I, Karlberg AC, Liljeholm M, Fraser AN, Madsen JE, Fjalestad T. Pegs not superior to screws for fixation of fractures of the proximal humerus. J Orthop Surg Res. 2022 Feb 2;17(1):66. doi: 10.1186/s13018-022-02947-3. PMID 35109905